CLINICAL TRIAL: NCT00277589
Title: TSH-adapted Therapy in a Large Randomized, Observer-blind, Placebo-controlled, Prospective Treatment Study of Patients With Nodular Goiter
Brief Title: LISA-study : Levothyroxin in Nodular Goiter
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: L_9133
Record Dates: First submitted 2006-01-13; First posted 2006-01-16 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-12

CONDITIONS: Goiter, Nodular
MeSH Terms: conditions — Goiter, Nodular | interventions — Iodides

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Levothyroxine-Na + iodide
- 2 (Active Comparator)
  Interventions: Drug: Levothyroxin-Na
- 3 (Active Comparator)
  Interventions: Drug: Iodide
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levothyroxin-Na — 1 tablet 30 minutes before breakfast
  Arms: 2
Drug: Levothyroxine-Na + iodide — 1 tablet 30 minutes before breakfast
  Arms: 1
Drug: Iodide — 1 tablet 30 minutes before breakfast
  Arms: 3
Drug: Placebo — 1 tablet 30 minutes before breakfast
  Arms: 4

SUMMARY:
Primary objective:

* To evaluate change in total volume of all nodules.

Secondary objectives:

* To evaluate change in goiter volume after a 12-months treatment, number of nodules and echogenicity of nodules.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Normal TSH value (target range between 0.6 - 3.0 mU/l)
* Thyroid nodules in a normal sized or enlarged thyroid at least one nodule (smaller/equal 20 % of volume with cystic change) with greater/equal 1.0 cm diameter, for nodules greater 1.0 cm the diagnosis must be performed according to the guideline for diagnostic standards of thyroid disorders.

Exclusion Criteria:

* Thyroid therapy within the last 3 years
* Known focal or diffuse structure autonomous thyroid
* Contraindication to iodine
* Concomitant treatment with iodine containing medication (i.e. amiodarone)
* Use of iodine-containing contrast medium within the last 6 weeks
* Presence of TPO antibodies (maximum two fold normal value)
* Symptomatic coronary heart disease
* Endocrine orbitopathy
* Known autoimmune thyreopathy
* Former radioiodine therapy or surgery
* Dermatitis herpetiformis
* Pathological laboratory results
* Participation in another clinical study with investigational medication within the last 30 days
* Pregnant or nursing female patients
* Female patients of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, unless they are surgically sterilized/hysterectomized or who are not using any other method considered sufficiently reliable by the investigator in individual cases.
* Severe or unstable cardiovascular diseases (e.g. severe angina pectoris, postmyocardial infarction syndrome and ventricular extrasystoles, symptomatic coronary heart disease), clinically relevant renal or hepatic diseases or disorders, any other clinically relevant condition that might enhance the risk for the study participant.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1024 (Actual)
Dates: Start 2004-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is to compare the change in total volume of all nodules after 12 months Levothyroxin treatment to the change after 12 months of each of the reference treatments (one of the two active controls or placebo) | after 12 months of treatment

SECONDARY OUTCOMES:
The change in goitre volume after Levothyroxin treatment will be compared to that after each reference treatment after 12 months treatment. | after 12 months treatment
Additionally, the change in the number of nodules after Levothyroxin treatment will be compared to each reference treatment after 12 months treatment. | after 12 months treatment
Echogenicity of the nodules after Levothyroxin treatment will be compared to each reference treatment after 12 months treatment. | after 12 months treatment

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Roscher, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Frankfurt, Germany